CLINICAL TRIAL: NCT05529719
Title: Effects of 12-Week Clinical Pilates Exercises in Young Adults With Mechanical Low Back Pain a Randomized Controlled Study
Brief Title: Effects of 12-Week Clinical Pilates Exercises on Mechanical Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Emir İbrahim IŞIK, Assistant Professor, Cukurova University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cp12wMlb
Record Dates: First submitted 2022-09-01; First posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Low Back Pain
Keywords: Clinical Pilates; Low back pain; Therapeutic Exercise
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial. Participants were randomly assigned to the intervention group and control group.
Masking Description: Due to the nature of the intervention, it was impossible to blind the participants and the researcher; however, we provided blinding during data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control group (Other): Patients assigned to the control group were given theoretical training and a brochure containing MBA information. The control group patients participating in the evaluation session were recommended to be included in the same clinical Pilates training conducted by the intervention group after the study was completed.
  Interventions: Other: Clinical Pilates Exercises

INTERVENTIONS:
Other: Clinical Pilates Exercises — Participants in the experimental group were included in the clinical Pilates intervention, which consisted of three weekly sessions for 50 minutes for 12 weeks. Clinical pilates sessions were performed by a clinically Pilates-certified instructor and a physiotherapist. The intervention was divided into three sections. Each session started with the warm-up section. The warm-up part started with breathing exercises, pelvic tilt centering, activation of deep trunk and pelvic floor muscles, and joint mobility. The Clinical Pilates exercises section consisted of matte level strength and flexibility exercises involving the trunk, upper and lower extremities. Finally, a cooling part was done that included some flexibility exercises.

SUMMARY:
Objective: This study evaluates the effect of 12-week clinical pilates exercises on young adults with mechanical low back pain.

Design: This is a randomized controlled trial. Setting: This study was conducted in a university's physiotherapy and exercise practice laboratory.

Cases: A total of 63 mechanical low back pain volunteers were included. Interventions: Participants were randomly assigned to the intervention group consisting of clinical Pilates exercises for 12 weeks (n = 31) or the control group not receiving any treatment (n = 32).

DETAILED DESCRIPTION:
Objective: This study evaluates the effect of 12-week clinical pilates exercises on young adults with mechanical low back pain.

Design: This is a randomized controlled trial. Setting: This study was conducted in a university's physiotherapy and exercise practice laboratory.

Cases: A total of 63 mechanical low back pain volunteers were included. The diagnosis of mechanical low back pain was made by a physical medicine and rehabilitation physician. Exercises are performed by an experienced physiotherapist with Clinical Pilates certification.

Interventions: Participants were randomly assigned to the intervention group consisting of clinical Pilates exercises for 12 weeks (n = 31) or the control group not receiving any treatment (n = 32).

Leading measures: Dysfunction was evaluated with the Oswestry Dysfunction Index. The Oswestry Disability Index (ODI)7,9 is the most commonly used outcome-measure questionnaire for low back pain in a hospital setting. Low bak pain was evaluated with the Visual Analog Scale (VAS). VAS is a tool used to help a person rate the intensity of certain sensations and feelings, such as pain. The visual analog scale for pain is a straight line with one end meaning no pain and the other end meaning the worst pain imaginable. And flexibility was evaluated with the sit and reach test test. The sit and reach test is a common measure of flexibility, and specifically measures the flexibility of the lower back and hamstring muscles. Measurements were performed at baseline and the end of the 12th week of the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 30 years of age; who had suffered from low back pain for at least three months; who had not used medication for low back pain in the last three months; who did not have a surgical history due to spinal problems; who did not have radiculopathy or other injuries such as fractures, stenosis or tumors in the spine; who had not received any treatment related to low back within the last six months; who had not previously continued pilates exercise; and who had sufficient physical autonomy to participate in the physical activities required by the study.

Exclusion Criteria:

* Volunteers who did not meet the inclusion criteria were excluded.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Prim Outcome - Oswestry Dysability Index | 12 weeks
  Pain-related functional competence was evaluated with the Oswestry disability index (ODI). ODI is a questionnaire consisting of 10 questions measuring the severity of pain, personal care, lifting, walking, sitting, standing, social life, sleep, travel status, and cognitive status of pain. Each question is evaluated between 0-5 points, and the ratio of the received score to the total answered question score gives the patient score. It is known that functional competence decreases and disability increases as the total score increases. It is interpreted as 0% to 20% - minimum disability 20% to 40% - moderate disability; 40% to 60% - severe disability; 60% to 80% - disabled 80% to 100% - bed-bound (or exaggerated symptoms).

SECONDARY OUTCOMES:
Sec Outcome - Visual Analogue Scale | 12 weeks
  Visual analog scale (VAS) scores were recorded to inquire about the pain status from the participants' registration information. In VAS, which is a horizontal line ten centimeters long, 0 indicates that there is no pain, while 10 indicates the most severe pain. Studies showed that VAS scores for those with chronic musculoskeletal pain corresponded to mild pain, 3.5 to 7.4 corresponded to moderate pain, and 7.5corresponds to severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Erkan KOZANOGLU, Professor, Study Chair — Cukurova University, Faculty of Medicine
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) of this study available to other researchers.
Supporting Information: Study Protocol
Time Frame: Timeless
Access Criteria: No individual participant data will be shared. Results will be published by the investigators in academic journals.

REFERENCES:
- [Background] Patrick N, Emanski E, Knaub MA. Acute and chronic low back pain. Med Clin North Am. 2014 Jul;98(4):777-89, xii. doi: 10.1016/j.mcna.2014.03.005. PMID 24994051
- [Background] Stoll J. THE LUMBAR SPINE: Mechanical Diagnosis and Therapy, R.A. Orthopedics. 1982 Oct;5(10):1378-82. doi: 10.3928/0147-7447-19821001-15. No abstract available. PMID 24830644
- [Background] Manchikanti L, Singh V, Falco FJ, Benyamin RM, Hirsch JA. Epidemiology of low back pain in adults. Neuromodulation. 2014 Oct;17 Suppl 2:3-10. doi: 10.1111/ner.12018. PMID 25395111
- [Background] van Tulder M, Malmivaara A, Esmail R, Koes B. Exercise therapy for low back pain: a systematic review within the framework of the cochrane collaboration back review group. Spine (Phila Pa 1976). 2000 Nov 1;25(21):2784-96. doi: 10.1097/00007632-200011010-00011. PMID 11064524
- [Background] Maher CG. Effective physical treatment for chronic low back pain. Orthop Clin North Am. 2004 Jan;35(1):57-64. doi: 10.1016/S0030-5898(03)00088-9. PMID 15062718
- [Background] Natour J, Cazotti Lde A, Ribeiro LH, Baptista AS, Jones A. Pilates improves pain, function and quality of life in patients with chronic low back pain: a randomized controlled trial. Clin Rehabil. 2015 Jan;29(1):59-68. doi: 10.1177/0269215514538981. Epub 2014 Jun 25. PMID 24965957